CLINICAL TRIAL: NCT06711744
Title: Effect of Time and Local Factors on Hydrophilic Tissue Level Implants in Post-extraction Sites: a RCT
Brief Title: ISQ Differences Between Different Implants in Post-extraction Sockets
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Paolo Carosi, Post-doctoral Researcher, University of Rome Tor Vergata
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: TLCVSTLX
Record Dates: First submitted 2024-11-21; First posted 2024-12-02 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-11

CONDITIONS: Bone Healing; Implant Stability

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TISSUE LEVEL X (Active Comparator): Implants with aggressive macro design
  Interventions: Diagnostic Test: Implant stability quotient
- TISSUE LEVEL C (Experimental): Implants with less aggressive macro design
  Interventions: Diagnostic Test: Implant stability quotient

INTERVENTIONS:
Diagnostic Test: Implant stability quotient — Screw a smart peg into the implant and record the values from a dedicated device

SUMMARY:
Two different implants will be used in post-extraction sockets and ISQ will be recorded monthly from insertion moment to 12 months of follow up to understand if ISQ can be affected by implant macro design

ELIGIBILITY:
Inclusion Criteria:

* Patients (at least 18 years old) presenting with failing tooth.
* no recession of gingival contour of tooth to be extracted
* no periodontal bone loss of neighboring teeth
* no implants in neighboring teeth
* class I extraction socket (intact buccal wall)
* atraumatic extraction of the tooth with intact socket walls remaining.

Exclusion Criteria:

* deep bite (severe II class)
* systemic disease (diabetes, osteoporosis)
* heavy smokers (more than 10 cigarettes/day)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
IMPLANT STABILITY QUOTIENT | Monthly from T0 (implant insertion) to T12 (12 months after implant placement)
  Values of risonance of implants taken by means of a dedicated device that translate the risonance of each implant into a number (0-99).

SECONDARY OUTCOMES:
Insertion torque | At implant placement
  Mechanical resistance of the bone at implant placement

CONTACTS AND LOCATIONS:
Locations (1):
- Paolo Carosi, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No